CLINICAL TRIAL: NCT06352970
Title: Effects of Tuberculosis Infection on Placental Development and Function
Brief Title: Effects of Tuberculosis Infection on Development and Function of the Placenta
Status: Recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Addis Ababa University (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Sponsor
Other Study IDs: LundU-2024
Record Dates: First submitted 2024-03-20; First posted 2024-04-08 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related; Tuberculosis Infection; Placenta Diseases
Keywords: placenta; tuberculosis; pregnancy complication
MeSH Terms: conditions — Latent Tuberculosis; Placenta Diseases; Tuberculosis; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Placenta tissue specimens Peripheral blood cell pellets Plasma aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women in labor: Women admitted to labor wards for delivery
  Interventions: Other: TB infection

INTERVENTIONS:
Other: TB infection — Outcomes will be compared with regard to result of interferon-gamma release assay test for TB infection

SUMMARY:
The goal of this observational study is to understand how tuberculosis (TB) infection impacts the function and development of the placenta, and whether TB infection can contribute to pregnancy-related disorders through effects on the placenta.

The main questions it aims to answer are:

* Does TB infection affect the structure of the placenta?
* Does TB infection affect the function of the placenta?

Pregnant women attending delivery clinics in Addis Abeba, Ethiopia, will be enrolled and classified for TB infection using a blood-based test. We will compare the following outcomes between women with TB infection and women without TB infection:

* Pathological lesions of the placenta
* Gene and protein expression patterns linked to pregnancy-related disorders
* Infant outcome at birth and at 6 weeks after birth

DETAILED DESCRIPTION:
Background:

Tuberculosis (TB) is an important cause of maternal morbidity and mortality globally, with the highest burden in low-income countries. Pregnancy has been associated with increased incidence of TB disease in register-based studies from Europe, suggesting that pregnancy can promote progression of TB infection (TBI). In a cohort of pregnant women living in Adama, a major Ethiopian city, one third of participants had TBI. Yet, the incidence of TB disease during pregnancy and post-partum follow-up in this cohort was relatively low (8 cases among 2000 participants during 4 years follow-up). Interestingly, levels of Mtb-triggered pro-inflammatory cytokines were elevated during later stages of pregnancy, suggesting increased bacterial activity during pregnancy in women with TBI. In addition, non-specific systemic inflammation markers in pregnant women with TBI were higher compared to pregnant women without TBI. It is likely that both these phenomena are due to pregnancy-induced immune modification of TB control.

The consequences of these immune changes in pregnancy have not been extensively studied. Apart from increased risk of progression to TB disease, it is possible that TBI in pregnant women could have other adverse health effects, in particular with regard to pregnancy outcome. In a recent register-based study of women living in Sweden with origin in TB-endemic countries screened for TBI in antenatal care, TBI was found to be associated with several types of adverse pregnancy outcomes. This finding suggests that TBI might affect development and function of the placenta, and could thus contribute to pregnancy complications. Several mechanisms can be involved in adverse effects of maternal infection on pregnancy outcome, including direct infection of fetal and/or placental tissue, as well as indirect effects mediated by systemic inflammation with impact on placental development and function.

This project is an in-depth study on the associations between TBI and TB disease and placental pathology, based on a cohort of women with delivery at Ethiopian public hospitals. The overall objective is to investigate placental pathology and markers of placental dysfunction in women with TB infection and TB disease, with correlation to Mtb immune responses and markers of mycobacterial activity and to characteristics of pregnancy disorders.

Project description Participants will be recruited and enrolled at labor wards at two public referral hospitals in Addis Abeba, Ethiopia. Study procedures will be performed by research nurses and research staff, as well as by trained regular staff based at the respective study sites. Study procedures will mainly be conducted during daytime during weekdays.

Study data will be obtained before as well as after delivery. Information from study participants will be collected using electronic structured questionnaires, including questions on socio-demographic condition, medical and obstetric history (current and previous pregnancies), as well as other variables recommended by the Global Pregnancy Collaboration COLLECT database. Detailed data on maternal and infant physical status (weight, height, mid-upper arm circumference, Apgar score), as well as delivery details, will be registered. Study data will be entered and uploaded using tablets connected to a REDCAP server. Blood samples for research purposes will be obtained in the labor ward before delivery. Before discharge from hospital, women will again be contacted by study staff for further information about the study. At this time, participants will also receive a scheduled date for the 6 week follow-up visit, as well as contact details for the study team.

Women with symptoms or signs suggestive of TB disease will be asked to submit two morning sputum samples for bacteriological TB investigations. Other investigations will be performed in women with suspected extrapulmonary TB (depending on the type of presentation; for example, fine needle aspiration in case of peripheral lymphadenopathy).

The whole placenta will be taken care of within 30 minutes after delivery by study pathology staff. First, the placenta will be characterized physically and macroscopically following a study protocol based on the recommendations of the Amsterdam Placental Workshop Group. The placenta will then be stored in formalin, with later embedment of selected parts in paraffin for histopathological investigations. In addition (from women with unlabored pregnancy who deliver at the TASH study site), portions of placenta tissue will be obtained for RNA and protein expression analyses, as well as for electron microscopy. These portions will be frozen on dry ice, with subsequent transfer to -80° C. Directly after delivery, cord blood will be collected in EDTA tubes (2-4 ml) for subsequent studies on RNA transcriptomic profile.

Venous blood will be collected in lithium heparin tubes (6 ml) for subsequent QuantiFERON TB-Plus (QFT) testing. In addition, blood will be collected in EDTA tubes (for antibody analyses; 4-6 ml).

QFT analysis for categorization of TBI status will be performed within one week after delivery. The result will be communicated to participants at the 6 week follow-up visit. In order to detect subclinical TB, women with TBI will be referred for chest X-ray (irrespective of symptoms) in connection with this visit. They will also be asked to submit two morning sputum samples for bacteriological TB analyses as described above.

Results from routine tests obtained at labor ward admission will be collected (HIV, malaria, syphilis, diabetes, renal function, liver function, blood count).

Laboratory methods

Mtb antigen-incubated blood:

Blood will be collected in lithium heparin tubes and separated into QFT tubes for incubation. Following incubation, blood will be centrifuged to separate supernatant from cell pellet. QFT ELISA will be performed according to the manufacturer's recommendation. Remaining supernatants will be stored in aliquots, and cell pellets will be separated and stored after addition of RNA-stabilizer. The Mtb-incubated cell pellet will be used for sequence-based analysis of RNA expression from selected women with TBI and TB disease to analyze mycobacterial activity patterns by comparison of patterns in women with TB infection and those with TB disease (including QFT-negative controls). Mtb-incubated supernatants will be analyzed for cytokines linked to TB activity (based on data from previous studies on TB immune dynamics during pregnancy), using Luminex technology platforms.

Unincubated blood:

Venous blood will be obtained in EDTA tubes for analysis of Mtb-specific antibodies.

Placenta:

Portions of placenta tissue will be obtained from different parts of macroscopically normal parts of the placenta. Portions will be obtained both for histopathological (formalin) and other studies (for freezer storage). All portions will be labelled with individual codes.

Methods for specific study aims:

1. To compare placental histopathology in women with and without TB infection/disease.

   For this aim, sections of paraffin-embedded placenta will be analyzed for different types of pathological changes. In addition, electron microscopy will be conducted from a subset of participants. Examinators will be blinded to TBI status and other characteristics of the participants. The histopathological changes will be scored. Subsequently, comparison with regard to TBI status will be performed to determine whether the occurrence of pathological changes differs between these categories, with adjustment for relevant concomitant conditions.
2. To compare RNA expression patterns in placenta tissue in women with and without TB infection/disease, and to correlate these findings with patterns associated with pregnancy disorders and placental dysfunction.

   For this aim, RNA expression patterns will be analyzed in placenta tissue from women with and without TB infection/disease, as well as from women with and without pre-defined pregnancy complications (pre-eclampsia, intra-uterine growth restriction). Participants for this study aim will be selected from the total cohort, based on TB infection/disease status. In order to avoid effects from labor, only participants with elective CS will be included for this analysis (unlabored placenta).

   Bulk sequencing will be used for analysis of RNA transcriptomics. Patterns of differentially expressed genes will be determined in these categories, with bioinformatic analysis on how differentially expressed genes from women with TB infection/disease correlate to those in women with pregnancy disorders (from the study population and from literature). These patterns will also be compared to individual pregnancy outcomes (adverse outcome, birth weight deviations).
3. To analyze protein expression in placenta tissue in pregnant women with and without TBI, and to correlate these patterns with placental pathology.

   For this aim, protein expression patterns in portions of unlabored placenta tissue will be characterized with regard to TB infection/disease status. Analysis will be done using mass spectrometry. The protein expression patterns found will subsequently be correlated to placental pathology and to pregnancy outcome characteristics.
4. To determine presence of Mtb in placental tissue in women with TBI. For this aim, participants with TB infection/disease will be included (along with a number of controls with negative QFT results). Portions of placental tissue will be investigated with methods to determine presence of Mtb, including immune histochemistry/in-situ hybridization techniques, and Mtb-specific probes that have been developed for use in paraffinized tissue samples.
5. To compare immune cell phenotypes in placental tissue in pregnant women with and without TB infection/disease, and to correlate these patterns with placental pathology.

   For this aim, paraffin-embedded placenta tissue will be used to identify immune cell phenotypes in women with regard to TBI status. Immunohistochemistry methods will be performed for this purpose.
6. To analyze Mtb-specific cytokine secretion and RNA expression patterns in Mtb-antigen-stimulated blood in women with TB infection/disease to delineate groups of women with different types of TB activity during pregnancy, and to correlate these patterns with placental findings.

   For this aim, women with TBI will be characterized with regard to immune profiles reflecting TB activity. These investigations will be based on Mtb-incubated supernatants and cell pellets, using Luminex techniques for analysis of Mtb-specific cytokines. RNA expression patterns will be analyzed using sequencing from selected participants (women with TBI, women with TB disease and QFT-negative women), followed by qPCR targeting differentially expressed genes from a larger number of women with TB infection/disease and QFT-negative women (in order to identify women with different types of TB infection, incipient and subclinical disease). The placental findings will be compared between these groups, with adjustment for other factors that may affect placental function and development.
7. To analyze TB-specific antibodies in lymphocyte supernatants in pregnant women with TBI to characterize mycobacterial activity and TB disease stage For this aim, BCG-specific antibodies will be analyzed in supernatants from cultured PBMCs from women with TBI. PBMCs will be isolated using cell preparation tubes, with culture on adapted media. Culture supernatants will be analyzed for presence of BCG-specific antibodies, and these patterns will be compared between participants to distinguish subsets of women with regard to active or incipient TB (with comparison of patterns in women with clinical TB disease and QFT-negative controls).

ELIGIBILITY:
Inclusion Criteria:

* Women admitted for delivery to study sites
* Written informed consent
* Age 18 years or greater

Exclusion Criteria:

* Chronic comorbidities (other than TB, HIV or pregnancy-related disorder)
* Twin pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with incipient delivery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of women with pathological placental findings according to the Amsterdam consensus criteria | 2025-2026
  Histopathological abnormalities linked to placental dysfunction and pregnancy-related disorders

SECONDARY OUTCOMES:
Proportions of women with placental RNA and protein expression patterns linked to pregnancy- related disorders | 2026-2027
  RNA and protein expression patterns in placenta linked to pregnancy-related disorders
Proportions of infants (born to participating women) with adverse outcome | 2025-2026
  Outcome of infants born to participants (at birth and 6 weeks after birth)

CONTACTS AND LOCATIONS:
Overall Officials: Per Bjorkman, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Gandhi Memorial Hospital, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.

REFERENCES:
- [Result] Sobhy S, Babiker Z, Zamora J, Khan KS, Kunst H. Maternal and perinatal mortality and morbidity associated with tuberculosis during pregnancy and the postpartum period: a systematic review and meta-analysis. BJOG. 2017 Apr;124(5):727-733. doi: 10.1111/1471-0528.14408. Epub 2016 Nov 11. PMID 27862893
- [Result] Jonsson J, Kuhlmann-Berenzon S, Berggren I, Bruchfeld J. Increased risk of active tuberculosis during pregnancy and postpartum: a register-based cohort study in Sweden. Eur Respir J. 2020 Mar 20;55(3):1901886. doi: 10.1183/13993003.01886-2019. Print 2020 Mar. PMID 31862768
- [Result] Zenner D, Kruijshaar ME, Andrews N, Abubakar I. Risk of tuberculosis in pregnancy: a national, primary care-based cohort and self-controlled case series study. Am J Respir Crit Care Med. 2012 Apr 1;185(7):779-84. doi: 10.1164/rccm.201106-1083OC. Epub 2011 Dec 8. PMID 22161161
- [Result] Walles J, Tesfaye F, Jansson M, Balcha TT, Sturegard E, Kefeni M, Merga G, Hansson SR, Winqvist N, Bjorkman P. Tuberculosis Infection in Women of Reproductive Age: A Cross-sectional Study at Antenatal Care Clinics in an Ethiopian City. Clin Infect Dis. 2021 Jul 15;73(2):203-210. doi: 10.1093/cid/ciaa561. PMID 32412638
- [Result] Tesfaye F, Walles J, Sturegard E, Winqvist N, Balcha TT, Kefeni M, Jansson M, Bjorkman P. Longitudinal Mycobacterium tuberculosis-Specific Interferon Gamma Responses in Ethiopian HIV-Negative Women during Pregnancy and Postpartum. J Clin Microbiol. 2021 Sep 20;59(10):e0086821. doi: 10.1128/JCM.00868-21. Epub 2021 Jul 28. PMID 34319803
- [Result] Tesfaye F, Sturegard E, Walles J, Bekele B, Bobosha K, Bjorkman P, Jansson M. Dynamics of Mycobacterium tuberculosis-Specific and Nonspecific Immune Responses in Women with Tuberculosis Infection during Pregnancy. Microbiol Spectr. 2022 Oct 26;10(5):e0117822. doi: 10.1128/spectrum.01178-22. Epub 2022 Aug 15. PMID 35969076
- [Result] Naik S, Alexander M, Kumar P, Kulkarni V, Deshpande P, Yadana S, Leu CS, Araujo-Pereira M, Andrade BB, Bhosale R, Babu S, Gupta A, Mathad JS, Shivakoti R. Systemic Inflammation in Pregnant Women With Latent Tuberculosis Infection. Front Immunol. 2021 Jan 27;11:587617. doi: 10.3389/fimmu.2020.587617. eCollection 2020. PMID 33584652
- [Result] Walles J, Winqvist N, Hansson SR, Sturegard E, Baqir H, Westman A, Kjerstadius T, Schon T, Bjorkman P. Pregnancy Outcomes in Women Screened for Tuberculosis Infection in Swedish Antenatal Care. Clin Infect Dis. 2024 Jan 25;78(1):125-132. doi: 10.1093/cid/ciad465. PMID 37572363
- [Result] Erez O, Romero R, Jung E, Chaemsaithong P, Bosco M, Suksai M, Gallo DM, Gotsch F. Preeclampsia and eclampsia: the conceptual evolution of a syndrome. Am J Obstet Gynecol. 2022 Feb;226(2S):S786-S803. doi: 10.1016/j.ajog.2021.12.001. PMID 35177220
- [Result] Myers JE, Myatt L, Roberts JM, Redman C; Global Pregnancy Collaboration (CoLab). COLLECT, a collaborative database for pregnancy and placental research studies worldwide. BJOG. 2019 Jan;126(1):8-10. doi: 10.1111/1471-0528.15393. Epub 2018 Aug 23. No abstract available. PMID 29978556
- [Result] Khong TY, Mooney EE, Ariel I, Balmus NC, Boyd TK, Brundler MA, Derricott H, Evans MJ, Faye-Petersen OM, Gillan JE, Heazell AE, Heller DS, Jacques SM, Keating S, Kelehan P, Maes A, McKay EM, Morgan TK, Nikkels PG, Parks WT, Redline RW, Scheimberg I, Schoots MH, Sebire NJ, Timmer A, Turowski G, van der Voorn JP, van Lijnschoten I, Gordijn SJ. Sampling and Definitions of Placental Lesions: Amsterdam Placental Workshop Group Consensus Statement. Arch Pathol Lab Med. 2016 Jul;140(7):698-713. doi: 10.5858/arpa.2015-0225-CC. Epub 2016 May 25. PMID 27223167
- [Result] Migliori GB, Ong CWM, Petrone L, D'Ambrosio L, Centis R, Goletti D. The definition of tuberculosis infection based on the spectrum of tuberculosis disease. Breathe (Sheff). 2021 Sep;17(3):210079. doi: 10.1183/20734735.0079-2021. PMID 35035549
- [Result] Ashenafi S, Aderaye G, Zewdie M, Raqib R, Bekele A, Magalhaes I, Lema B, Habtamu M, Rekha RS, Aseffa G, Maeurer M, Aseffa A, Svensson M, Andersson J, Brighenti S. BCG-specific IgG-secreting peripheral plasmablasts as a potential biomarker of active tuberculosis in HIV negative and HIV positive patients. Thorax. 2013 Mar;68(3):269-76. doi: 10.1136/thoraxjnl-2012-201817. Epub 2012 Aug 24. PMID 22923457
- [Result] Mathad JS, Yadav S, Vaidyanathan A, Gupta A, LaCourse SM. Tuberculosis Infection in Pregnant People: Current Practices and Research Priorities. Pathogens. 2022 Dec 6;11(12):1481. doi: 10.3390/pathogens11121481. PMID 36558815